CLINICAL TRIAL: NCT02605733
Title: The Neu-Prem Trial: Neuromonitoring of Preterm Newborn Brain During Birth Resuscitation
Acronym: Neu-Prem
Status: Completed | Type: Observational
Sponsor: Sharp HealthCare (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research, Sharp HealthCare
Other Study IDs: Neu-Prem
Record Dates: First submitted 2015-10-30; First posted 2015-11-16 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Neurologic Manifestations; Premature Birth; Hypoxia-Ischemia, Brain
Keywords: Premature infant; Amplitude integrated EEG; Near-infrared spectroscopy
MeSH Terms: conditions — Neurologic Manifestations; Premature Birth; Hypoxia-Ischemia, Brain | interventions — Electroencephalography; Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EEG — amplitude integrated electroencephalography
  Other Names: amplitude integrated electroencephalography
Device: NIRS — regional tissue oximetry
  Other Names: Near-infrared spectroscopy

SUMMARY:
The purpose of this study is to characterize the normal brain function of premature infants (23 to 31+6 weeks GA) during birth transition and through the first 72 hours of life.

DETAILED DESCRIPTION:
The investigators will measure components of brain function using two sophisticated, non-invasive technologies. First, amplitude integrated electroencephalography (EEG), a "simplified" EEG with four sensors (single channel), enables continuous non-invasive monitoring of cerebral activity. Second, near-infrared spectroscopy (NIRS) is another non-invasive technology that allows continuous real-time measurement of regional tissue oxygen utilization of the brain. Both technologies have been used in newborns and have been predictive of brain injury or neurodevelopmental impairment.

ELIGIBILITY:
Inclusion Criteria:

* 23 to 31+6 weeks gestational age at birth

Exclusion Criteria:

* Known congenital anomalies
* Parents refuse consent
* Neonatologist declined due to subject instability

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants delivered at 23 to 31 +6 weeks gestational age at Sharp MBHWN.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12-31 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
EEG | Birth to 72 hours of life
  amplitude integrated EEG to measure brain activity
NIRS | Birth to 72 hours of life
  Cerebral tissue oxygen saturation (StO2), Near-infrared spectroscopy to measure brain perfusion

SECONDARY OUTCOMES:
Apgar scores | 1, 5 and 10 minutes of life if applicable
  1 and 5 minute Apgar scores
Cord gases | Upon delivery
  Arterial or venous pH (acid/base), base deficit
Resuscitation intervention | From birth to 10 minutes of life
  Fraction of inspired oxygen (FiO2), cpap, positive pressure ventilation (PPV), intubations.
Maximum FiO2 | From birth to 10 minutes of life
  Maximum FiO2 during resuscitation at birth
Maximum peak inspiratory pressure | From birth to 10 minutes of life
  Peak inspiratory pressure of respiratory support
Heart rate | Birth to 72 hours of life
Heart rate by EKG during resuscitation (substudy) | Birth
  A substudy of 40 infants will have EKG leads placed on newborns during resuscitation; 20 will have the display blinded, and 20 will have values available to the team. The amount of resuscitation (mean airway pressure FiO2 will be compared between groups).
Cardiac output | From neonatal intensive care unit (NICU) admission through 72 hours of life
Mean arterial blood pressure | From NICU admission through 72 hours of life
Use of cardiac inotropes | From birth through discharge to home, up to 9 months of age
  Dopamine, dobutamine, epinephrine
Head Ultrasound | Within 24 hours of life and at approximately 72 hours of life
  Cranial ultrasonography
MRI | From birth through discharge to home, up to 9 months of age
  Presence of brain injury (e.g. intraventricular hemorrhage (IVH), (PVL)
Neurodevelopmental impairment at 2 year follow up | 18 to 30 months corrected gestational age
  Neurodevelopmental assessment at 2 year corrected gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

REFERENCES:
- [Background] Peng S, Boudes E, Tan X, Saint-Martin C, Shevell M, Wintermark P. Does near-infrared spectroscopy identify asphyxiated newborns at risk of developing brain injury during hypothermia treatment? Am J Perinatol. 2015 May;32(6):555-64. doi: 10.1055/s-0034-1396692. Epub 2015 Jan 16. PMID 25594221
- [Background] Ancora G, Maranella E, Locatelli C, Pierantoni L, Faldella G. Changes in cerebral hemodynamics and amplitude integrated EEG in an asphyxiated newborn during and after cool cap treatment. Brain Dev. 2009 Jun;31(6):442-4. doi: 10.1016/j.braindev.2008.06.003. Epub 2008 Jul 22. PMID 18650042
- [Background] Ancora G, Maranella E, Grandi S, Sbravati F, Coccolini E, Savini S, Faldella G. Early predictors of short term neurodevelopmental outcome in asphyxiated cooled infants. A combined brain amplitude integrated electroencephalography and near infrared spectroscopy study. Brain Dev. 2013 Jan;35(1):26-31. doi: 10.1016/j.braindev.2011.09.008. Epub 2011 Nov 13. PMID 22082686
- [Background] Gucuyener K, Beken S, Ergenekon E, Soysal S, Hirfanoglu I, Turan O, Unal S, Altuntas N, Kazanci E, Kulali F, Koc E, Turkyilmaz C, Onal E, Atalay Y. Use of amplitude-integrated electroencephalography (aEEG) and near infrared spectroscopy findings in neonates with asphyxia during selective head cooling. Brain Dev. 2012 Apr;34(4):280-6. doi: 10.1016/j.braindev.2011.06.005. Epub 2011 Jul 7. PMID 21741190
- [Background] Toet MC, Lemmers PM. Brain monitoring in neonates. Early Hum Dev. 2009 Feb;85(2):77-84. doi: 10.1016/j.earlhumdev.2008.11.007. Epub 2009 Jan 17. PMID 19150756
- [Background] Tao JD, Mathur AM. Using amplitude-integrated EEG in neonatal intensive care. J Perinatol. 2010 Oct;30 Suppl:S73-81. doi: 10.1038/jp.2010.93. PMID 20877412
- [Background] Fuchs H, Lindner W, Buschko A, Almazam M, Hummler HD, Schmid MB. Brain oxygenation monitoring during neonatal resuscitation of very low birth weight infants. J Perinatol. 2012 May;32(5):356-62. doi: 10.1038/jp.2011.110. Epub 2011 Aug 18. PMID 21852771
- [Background] Katheria AC, Leone TA, Woelkers D, Garey DM, Rich W, Finer NN. The effects of umbilical cord milking on hemodynamics and neonatal outcomes in premature neonates. J Pediatr. 2014 May;164(5):1045-1050.e1. doi: 10.1016/j.jpeds.2014.01.024. Epub 2014 Feb 20. PMID 24560179
- [Background] Katheria A, Blank D, Rich W, Finer N. Umbilical cord milking improves transition in premature infants at birth. PLoS One. 2014 Apr 7;9(4):e94085. doi: 10.1371/journal.pone.0094085. eCollection 2014. PMID 24709780
- [Background] Noori S, McCoy M, Anderson MP, Ramji F, Seri I. Changes in cardiac function and cerebral blood flow in relation to peri/intraventricular hemorrhage in extremely preterm infants. J Pediatr. 2014 Feb;164(2):264-70.e1-3. doi: 10.1016/j.jpeds.2013.09.045. Epub 2013 Oct 30. PMID 24183212
- [Background] Zhang Y, Chan GS, Tracy MB, Lee QY, Hinder M, Savkin AV, Lovell NH. Cerebral near-infrared spectroscopy analysis in preterm infants with intraventricular hemorrhage. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:1937-40. doi: 10.1109/IEMBS.2011.6090547. PMID 22254711
- [Background] Song J, Zhu C, Xu F, Guo J, Zhang Y. Predictive value of early amplitude-integrated electroencephalography for later diagnosed cerebral white matter damage in preterm infants. Neuropediatrics. 2014 Oct;45(5):314-20. doi: 10.1055/s-0034-1382823. Epub 2014 Jul 8. PMID 25003781
- [Background] Benders MJ, Palmu K, Menache C, Borradori-Tolsa C, Lazeyras F, Sizonenko S, Dubois J, Vanhatalo S, Huppi PS. Early Brain Activity Relates to Subsequent Brain Growth in Premature Infants. Cereb Cortex. 2015 Sep;25(9):3014-24. doi: 10.1093/cercor/bhu097. Epub 2014 May 27. PMID 24867393
- [Background] Pichler G, Avian A, Binder C, Zotter H, Schmolzer GM, Morris N, Muller W, Urlesberger B. aEEG and NIRS during transition and resuscitation after birth: promising additional tools; an observational study. Resuscitation. 2013 Jul;84(7):974-8. doi: 10.1016/j.resuscitation.2012.12.025. Epub 2013 Jan 8. PMID 23313424
- [Derived] Katheria AC, Harbert MJ, Nagaraj SB, Arnell K, Poeltler DM, Brown MK, Rich W, Hassen KO, Finer N. The Neu-Prem Trial: Neuromonitoring of Brains of Infants Born Preterm During Resuscitation-A Prospective Observational Cohort Study. J Pediatr. 2018 Jul;198:209-213.e3. doi: 10.1016/j.jpeds.2018.02.065. Epub 2018 Apr 18. PMID 29680471